CLINICAL TRIAL: NCT02355184
Title: Extension of Protocol PRO140_CD01 to Further Evaluate Long-term Suppression of HIV-1 Replication Following Substitution of Stable Combination ART With PRO 140 (Monoclonal CCR5 Antibody) Monotherapy in Adult Subjects With HIV-1 Infection
Brief Title: An Extension of Protocol PRO 140_CD01 Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA required the sponsor to halt enrollment in the trial and transition participants to available therapies for the treatment of their disease. The trial was subsequently terminated once participants were transitioned.
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 140_CD 01-Extension
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: HIV; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — leronlimab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRO 140 (Experimental): PRO 140 350mg weekly subcutaneous (SC) injection.
  Interventions: Drug: PRO 140 350mg weekly subcutaneous (SC) injection.

INTERVENTIONS:
Drug: PRO 140 350mg weekly subcutaneous (SC) injection. — CCR5 Antagonist
  Other Names: PRO 140

SUMMARY:
This is an extension of Protocol PRO 140_CD 01 to further evaluate the long-term suppression of HIV-1 replication following substitution of stable combination antiretroviral therapy with a PRO 140 (Monoclonal CCR5 antibody) monotherapy in adult subjects with HIV-1 infection

DETAILED DESCRIPTION:
This study is a Phase 2b, multi-center, extension study designed to evaluate the long-term efficacy, safety, and tolerability of PRO 140 monotherapy for the maintenance of viral suppression in patients who were stable on combination antiretroviral therapy and completed 12 weeks of treatment under PRO 140_CD 01 Treatment Substitution Study without experiencing virologic failure.

Consenting patients will continue to receive PRO 140 monotherapy until investigational product (IP) receives marketing approval or investigational new drug (IND) is withdrawn by Sponsor. There is one week overlap of existing retroviral regimen and PRO 140 at the end of the treatment extension phase in subjects who do not experience virologic failure.

PRO 140 will be administered as a 350 mg subcutaneous injection weekly during treatment extension phase. Study participants will be monitored for viral rebound on a weekly basis following initiation of PRO 140 monotherapy and will re-initiate their previous antiretroviral regimen if plasma HIV-1 RNA levels rise above 400 copies/ml on two consecutive blood draws at least 3 days apart.

.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed 12 weeks of treatment in PRO 140_CD01 study without experiencing virologic failure.
2. Both male and female patients and their partners of childbearing potential must agree to use appropriate birth control methods (birth control pills, barriers, or abstinence) throughout the study duration (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative urine pregnancy test prior to receiving the first dose of study drug.
3. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria:

1. Not currently enrolled in PRO140_CD01 Treatment Substitution Study
2. Any acquired immune deficiency syndrome (AIDS)-defining illness according to the 1993 Centers for Disease Control and Prevention (CDC) AIDS surveillance definition
3. Laboratory test values ≥ grade 4 DAIDS laboratory abnormality.
4. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
5. Unexplained temperature >38.5C (101.3F) for seven consecutive days within 14 days prior to the first study dose
6. Diagnosed with either substance dependence or substance abuse or any history of a concomitant condition (e.g., medical, psychologic, or psychiatric) that in the opinion of the primary care provider and/or site investigator would interfere with the subject's successful completion of the study requirements
7. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Principal Investigator — CytoDyn, Inc.
Locations (1):
- CD01-Extension Investigational Site, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang XL, Reed JS, Webb GM, Wu HL, Le J, Bateman KB, Greene JM, Pessoa C, Waytashek C, Weber WC, Hwang J, Fischer M, Moats C, Shiel O, Bochart RM, Crank H, Siess D, Giobbi T, Torgerson J, Agnor R, Gao L, Dhody K, Lalezari JP, Bandar IS, Carnate AM, Pang AS, Corley MJ, Kelly S, Pourhassan N, Smedley J, Bimber BN, Hansen SG, Ndhlovu LC, Sacha JB. Suppression of human and simian immunodeficiency virus replication with the CCR5-specific antibody Leronlimab in two species. PLoS Pathog. 2022 Mar 31;18(3):e1010396. doi: 10.1371/journal.ppat.1010396. eCollection 2022 Mar. PMID 35358290

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO 140: PRO 140 350mg weekly SC injection.
  PRO 140 350mg weekly SC injection.: C-C chemokine receptor type 5 (CCR5) Antagonist
Period: Overall Study
Arm/Group | PRO 140
Started | 20
Completed | 8
Not Completed | 12
Not completed — Lost to Follow-up | 2
Not completed — Study Terminated | 10

BASELINE CHARACTERISTICS:
Population: Subjects with HIV-1 infection who did not experience virologic failure while in the treatment phase of the PRO 140_CD 01 study.
Groups:
- PRO 140: PRO 140 350mg weekly SQ (subcutaneous) injection.
  PRO 140 350mg weekly SQ injection.: CCR5 Antagonist
Arm/Group | PRO 140
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 56.05 [32 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20
Time since HIV Diagnosis [Mean (Full Range); unit: years] — Time in years since HIV original diagnosis taken at visit 1
  years | 10 [2 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Time to Virologic Failure After Initiating PRO 140 Monotherapy
Description: Virologic failure (VF) is defined as two consecutive HIV-1 RNA levels of ≥ 400 copies/ml separated by at least 3 days. The time to VF will be compared to a historical data (i.e., time to HIV-1 RNA viral load > 500 copies/mL of 29 days). The statistical comparison will be conducted using Wilcoxon rank sum test and the median time to Virologic Failure for this study will be compared to 30 days.
Time Frame: From treatment extension visit 1 (TE1) until virologic failure, assessed up to 125 weeks.
Population: The efficacy population consists of all subjects who received at least one dose of leronlimab (PRO 140).
Measure: Mean (Standard Deviation); unit: days
Groups:
- PRO 140: PRO 140 350mg weekly SQ injection.
Arm/Group | PRO 140
Number analyzed (Participants) | 20
days | 228.8 (225.6)

2. Secondary Outcome: Proportion of Participants With Virologic Failure After Initiating PRO 140 Monotherapy.
Description: Virologic failure is defined as two consecutive HIV-1 RNA levels of ≥ 400 copies/ml separated by at least 3 days.
Time Frame: From treatment extension visit 1 (TE1) until virologic failure, assessed up to 125 weeks.
Population: The efficacy population consists of all subjects who received at least one dose of leronlimab (PRO 140).
Measure: Number; unit: proportion of participants
Groups:
- PRO 140: PRO 140 350mg weekly SQ injection.
  PRO 140 350mg weekly SQ injection.: CCR5 Antagonist
Arm/Group | PRO 140
Number analyzed (Participants) | 20
proportion of participants | 0.3

3. Secondary Outcome: Mean Change in Viral Load (HIV-1 RNA Levels)
Description: Mean change from baseline of HIV-1 RNA levels was assessed for each week during the treatment phase up until week 58. Weighted mean change in viral load (HIV-1 RNA levels) were calculated from baseline to week 58.
Time Frame: From treatment extension visit TE2 (defined as baseline), until week 58 of extension treatment.
Population: The efficacy population consists of all subjects who received at least one dose of leronlimab (PRO 140). Baseline was defined as TE2. Any subjects with an undefined change from baseline due to missing data were excluded. The following imputations were used in the statistical analysis: "<40" copies/mL as 40 "Target not detected" as 20.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | PRO 140
Number analyzed (Participants) | 16
copies/mL | 147.34 (263.60)

4. Secondary Outcome: Mean Change in CD4 Cell Count
Description: Mean change in CD4 cell count from baseline (TE2 visit) was assessed for each week during the treatment phase up until week 58. The average mean change was calculated from baseline to week 58.
Time Frame: From treatment extension visit TE2 (defined as baseline), until week 58 of extension treatment.
Population: The efficacy population consists of all subjects who received at least one dose of leronlimab (PRO 140). Baseline was defined as TE2. Any subjects with an undefined change from baseline due to missing data were excluded.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | PRO 140
Number analyzed (Participants) | 16
cells/uL | 22 (111)

5. Secondary Outcome: Change in Quality of Life Metrics (up to TE107)
Description: A Quality of Life (QoL) assessment using ACTG SF-21 was planned to be performed at screening visit (SV1), once every four weeks from treatment visit 4 (TE4) through treatment visit 107 (TE107), and at end of treatment (EOT). The ACTG SF-21 has 8 QoL domains with a standard score ranging from 0 (worst) to 100 (best).
Time Frame: From TE4 (baseline) through every fourth weekly visits to treatment visit 107 (TE107) or EOT, up to 125 weeks.
Population: No QoL data was collected at screening visit (SV1) for any of the participants. For 5 participants Quality-of-life (QoL) results were either not collected or they had undefined change from baseline due to missing data.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | PRO 140
Number analyzed (Participants) | 15
score | 1.4 (5.9)

6. Other Pre Specified Outcome: Tolerability of Repeated Subcutaneous Administration of PRO 140 as Assessed by Study Participants(Using Visual Analogue Scale) and by Investigator-evaluation of Injection Site Reactions.
Description: Tolerability of repeated subcutaneous administration of PRO 140 was planned to be assessed by the study participants using a Visual Analogue Scale, and by investigator-evaluation of injection site reactions. Injection site reaction assessment was not completed when subjects performed self-administration.
Time Frame: From TE1 (first treatment administration) weekly until last treatment visit (up to 125 weeks)
Population: Data on tolerability of repeated subcutaneous (SC) administration of PRO 140 was not collected.
Arm/Group | PRO 140
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Number of Participants With Grade 3 or 4 Adverse Events as Defined by the DAIDS Adverse Event Scale
Description: The Division of AIDS (DAIDS) grading table provides an adverse event severity grading scale ranging from grades 1 to 5 with descriptions for each adverse event based on the following general guidelines:
  * Grade 1 indicates a mild event
  * Grade 2 indicates a moderate event
  * Grade 3 indicates a severe event
  * Grade 4 indicates a potentially life-threatening event
  * Grade 5 indicates death (Note: This grade is not specifically listed on each page of the grading table).
Time Frame: From the first treatment visit (TE1) until final study visit, up to a 125 weeks.
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140
Number analyzed (Participants) | 20
Participants | 7

8. Other Pre Specified Outcome: Number of Participants With at Least One Treatment-related Serious Adverse Event.
Description: Treatment-related serious adverse events are defined as serious events with an onset on or after the first treatment.
  A serious adverse event is defined as any adverse event that:
  * Results in death
  * Is life threatening (the subject is at immediate risk of dying from the AE)
  * Requires subject hospitalization or prolongs existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: From the first treatment visit (TE1) until final study visit up to 125 weeks.
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of the first treatment and continued up until the final study visit to evaluate safety of PRO140 (up to a maximum of 91 months).
Arm/Group | PRO 140
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO 140 (N=20)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (3)
Syncope (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO 140 (N=20)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Epididymitis (Infections and infestations) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Abscess limb (Infections and infestations) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chills (General disorders) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dissociation (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Drug Abuse (Psychiatric disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (4)
Gastrooeophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Giardiasis (Infections and infestations) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hyporeflexia (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3)
Malaise (General disorders) | 1 (1)
Migrane (Nervous system disorders) | 1 (1)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Oral Candidiasis (Infections and infestations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pustule (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Shigella infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (6)
Substance abuse (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syphillis (Infections and infestations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (7)
Vaccination site rash (General disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Certain lab data were not collected or were otherwise unavailable for analysis or reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02355184/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02355184/SAP_001.pdf